CLINICAL TRIAL: NCT01334255
Title: A Phase 1b Multi-Center, Open-Label and Randomized Study of iSONEP (Sonepcizumab/LT1009) Administered as Intravitreous Injections to Subjects With PED Secondary to Exudative Age-Related Macular Degeneration or Polypoidal Choroidal Vasculopathy
Brief Title: iSONEP to Treat Persistent Pigment Epithelial Detachment (PED) in Subjects With Exudative Age-Related Macular Degeneration (AMD) or Polypoidal Choroidal Vasculopathy (PCV)
Acronym: PED
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision; not safety related
Sponsor: Lpath, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT1009-Oph-002
Record Dates: First submitted 2011-04-08; First posted 2011-04-13 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2012-01

CONDITIONS: Pigment Epithelial Detachment
Keywords: Pigment epithelial detachment; Exudative age-related macular degeneration; Polypoidal choroidal vasculopathy
MeSH Terms: conditions — Retinal Detachment; Polypoidal Choroidal Vasculopathy | interventions — sonepcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 mg of iSONEP (sonepcizumab/LT1009) (Experimental): iSONEP (sonepcizumab/LT1009) is a humanized murine monoclonal antibody to sphingosine 1-phosphate
  Interventions: Drug: iSONEP (sonepcizumab/LT1009)
- 2.0 mg of iSONEP (sonepcizumab/LT1009) (Experimental): iSONEP (sonepcizumab/LT1009) is a humanized murine monoclonal antibody to sphingosine 1-phosphate
  Interventions: Drug: iSONEP (sonepcizumab/LT1009)

INTERVENTIONS:
Drug: iSONEP (sonepcizumab/LT1009) — Up to 3 doses of iSONEP given monthly will be administered as intravitreous injections in the ophthalmologist's office.

SUMMARY:
LT1009-Oph-002 is a Phase 1b study designed to evaluate the safety and potential efficacy of iSONEP following one, two or three injections of iSONEP, as needed, for the treatment of Pigment Epithelial Detachment (PED) secondary to PED Secondary to Exudative Age-Related Macular Degeneration (AMD) or Polypoidal Choroidal Vasculopathy (PCV).

DETAILED DESCRIPTION:
Sixteen (16) subjects per dose group who have received a minimum of 3 and no more than 7 doses of an anti-VEGF agent (i.e., Lucentis or Avastin), and whose PED has not decreased by greater than 25% in height despite therapy, will be enrolled for a total of 32 subjects. The presence of PED diagnosed by the Investigator will be confirmed by SDOCT, ICG and FA by a digital imaging reading center prior to subject enrollment. The ability of iSONEP to induce regression of persistent PED in subjects with exudative AMD or PCV despite previous treatment with an anti-VEGF agent will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 50 years of age with a diagnosis of PED secondary to AMD or PCV
* Serous and/or fibrovascular PED secondary to exudative AMD or secondary to PCV (confirmed by SDOCT, FA and ICG) that has not demonstrated at least a 25% decrease in the height of the PED (from the onset of anti-VEGF therapy) following a minimum of 3 doses of an anti-VEGF agent (i.e., Lucentis or Avastin)
* PED that has a height greater than 100 μm
* Presence of CNV secondary to (i) AMD (based on FA) or (ii) PCV (based on ICG)
* ETDRS BCVA of 20/32 to 20/320 (letter score of 73 to 25) in the study eye
* ETDRS visual acuity of 20/400 or better in the fellow eye

Exclusion Criteria:

* Subjects previously treated with, or are currently receiving treatment with another investigational agent or device for neovascular AMD in the study eye
* Subjects who have received < 3 and > 7 anti-VEGF treatments in the study eye
* Subjects with retinal angiomatous proliferation (RAP lesion)
* Lucentis or Avastin within 30 days prior to Day 1 in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability following one, two or three intravitreous injections of iSONEP | 8 months
  The number of participants with adverse events; changes in electrocardiogram parameters, diastolic and systolic blood pressure, pulse, temperature and intraocular pressure from baseline to the end of the study.

SECONDARY OUTCOMES:
To evaluate various efficacy outcomes throughout the study | 8 months
  * Changes in subretinal and intraretinal fluid, in retinal thickness and in size and height of PED compared with baseline at Days 30, 45, 60 and 90
  * Changes in CNV lesion area from baseline
  * Time course to regression of PED; proportion of subjects with complete resolution of PED following a single, second or third IVT iSONEP injection
  * Changes in VA; proportion of eyes gaining > or = 0, 5, 10 and 15 letters on ETDRS
  * Proportion of subjects with an improvement from baseline in VFQ-25 overall composite score to Day 60, Month 4 and Month 8
  * Time to re-treatment with anti-VEGF therapy
To evaluate the immunogenicity (antibody response) of iSONEP following multiple intravitreous injections | 8 months
  Production and/or changes in antibody concentration to iSONEP from baseline to the end of the study
To characterize the systemic pharmacokinetic profile of iSONEP | 8 months
  For the 2.0 mg dose of iSONEP
  * Maximum plasma concentration
  * Area under the concentration versus time curve
  * Terminal half-life
  * Terminal elimination constant
  * Time of maximum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Stoller, MD, Study Chair — Lpath, Inc.
Locations (5):
- United States (5):
  - Center For Retina & Macular Disease, Winter Haven, Florida
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, Austin, Texas